CLINICAL TRIAL: NCT00549120
Title: A Study to Optimise the Propranolol Block Model for Assessment of the Pharmacological Activity of Bronchodilators in Healthy Volunteers.
Brief Title: Optimising the Propranolol Block Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MAB104954
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Healthy Subjects; muscarinic receptor antagonist; propranolol; beta-blocker; beta-agonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Propranolol; Albuterol; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Propranolol alone (Experimental): Propranolol 80 mg (5 doses at 6 hourly intervals)
  Interventions: Drug: Propranolol
- Propranolol + salbutamol (Experimental): Propranolol 80 mg (5 doses at 6 hourly intervals) + salbutamol 600 μg (4 doses at 6 hourly intervals)
  Interventions: Drug: Propranolol; Drug: Salbutamol
- Salbutamol alone (Experimental): Salbutamol 600 μg (4 doses at 6 hourly) + placebo (5 doses at 6 hourly intervals)
  Interventions: Drug: Salbutamol; Drug: Placebo
- Placebo (Placebo Comparator): Placebo (5 doses at 6 hourly)
  Interventions: Drug: Placebo
- Propranolol + ipratropium + salbutamol (Experimental): Propranolol 80 mg (2 doses at 6 hourly intervals) + ipratropium bromide 40 μg (2 doses at 6 hourly interval) + salbutamol 600 μg (1 dose)
  Interventions: Drug: Propranolol; Drug: Salbutamol; Drug: Ipratropium
- Placebo + ipratropium + salbutamol (Experimental): Placebo (2 doses at 6 hourly intervals) + ipratropium bromide 40 μg (2 doses at 6 hourly interval) + salbutamol 600 μg (1 dose)
  Interventions: Drug: Salbutamol; Drug: Ipratropium; Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — 40 mg tablets
  Arms: Propranolol + ipratropium + salbutamol; Propranolol + salbutamol; Propranolol alone
Drug: Salbutamol — Metered dose inhaler (600 μg)
  Arms: Placebo + ipratropium + salbutamol; Propranolol + ipratropium + salbutamol; Propranolol + salbutamol; Salbutamol alone
Drug: Ipratropium — Metered dose inhaler (40 μg)
  Arms: Placebo + ipratropium + salbutamol; Propranolol + ipratropium + salbutamol
Drug: Placebo — Placebo for propranolol tablets
  Arms: Placebo; Placebo + ipratropium + salbutamol; Salbutamol alone

SUMMARY:
Optimising the propranolol block model

DETAILED DESCRIPTION:
The bronchodilatory effects of inhaled beta2 agonists and anti-muscarinic drugs are the mainstay of symptomatic treatment of asthma and Chronic Obstructive Pulmonary Disease (COPD). A new approach is to combine both pharmacological approaches in a single molecule - ie a dual pharmacophore. It will be necessary to explore the relative contribution of the beta2 agonist versus anti-muscarinic bronchodilator properties of such a molecule. One way to do that is to block one of the components. Inhibition of beta2 agonist-mediated bronchodilatation by the non-selective beta-blocker propranolol is an established experimental method. Therefore this method may be useful in exploring the pharmacology of a dual pharmacophore.

Published studies have generally looked at the effect of a single dose of propranolol on a beta2 agonist over a relatively short period of time (a few hours). There is a desire to develop long acting bronchodilators that require once daily dosing only. Thus any dual pharmacophore developed is likely to have 24 hour duration of action after a single dose. Therefore to use this method of beta blockade to inhibit beta2 agonist mediated bronchodilation, it is necessary to confirm a dosing regimen of propranolol that has acceptable tolerability and is effective in blocking the effects of a beta2 agonist over 24 hours. That is the main purpose of this study.

It is also important to confirm that the bronchodilator effect of an antimuscarinic is unaffected by beta blockade. In addition, it is of interest to examine the bronchodilator effect of a combination of an antimuscarinic and beta2 agonist in healthy volunteers and the effect of propranolol on the combination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female aged between 18 and 50 years.
* Body mass index within the range 19-29.9 kilograms/metre2
* Forced Expiratory Volume in 1 second (FEV1) >80% predicted and a FEV1/ Forced Vital Capacity (FVC) ratio > 0.7
* The subject has an increase in sGAW of >% over pre-dose baseline within 2 h of administration of 400 ug salbutamol by MDI inhaler at screening or in the 3 months before screening.
* Subject has an increase in sGaw of 25% over pre-dose baseline within 2 h following 40 ug ipratropium bromide at screening or in the 3 months before screening
* Subjects are current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of < 10 pack years.

Exclusion criteria:

* A past or present disease, which as judged by the Investigator and medical monitor may affect the outcome of the study or the safety of the subject
* History of respiratory disease
* Significant abnormal 12 lead ECG, QTc(B) and QTc(F) value at screening >450msec on an individual ECG or a PR interval outside the range 120-210 msec
* Supine mean heart rate outside the range 45-90 beats per minute (bpm) at screening
* Subject has donated a unit of blood within the 56 days or intends to donate within 56 days after completing the study
* Subject is currently taking regular (or course of) medication whether prescribed or not (with the exception of contraceptives, including vitamins and herbal remedies such as St John's Wort)
* Subject has participated in a clinical study with a New Chemical Entity (NCE) within the past 1 month
* Infected with the Hepatitis B, Hepatitis C, or HIV virus
* Subject has a history of drug or other allergy, which, in the opinion of the Investigator, contraindicates their participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-08-15 (Actual); Primary Completion 2007-10-26 (Actual); Study Completion 2007-10-26 (Actual)

PRIMARY OUTCOMES:
Specific airway conductance (sGAW) | Pre-dose and up to 26 h post-dose

SECONDARY OUTCOMES:
Tolerability: adverse events, 12 lead ECG, blood pressure and heart rate | Study duration
Propranolol pharmacokinetics | Pre-dose and up to 28 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study MAB104954 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/MAB104954?search=study&search_terms=104954#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: MAB104954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: MAB104954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: MAB104954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: MAB104954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: MAB104954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: MAB104954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: MAB104954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register